CLINICAL TRIAL: NCT00801619
Title: Bilicurves: Using Information Technology to Integrate Clinical Practice Guidelines Into the Management of Neonatal Hyperbilirubinemia
Brief Title: Bilicurves: Using Information Technology to Improve the Management of Neonatal Hyperbilirubinemia
Status: Completed | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, John Patrick Co, Principal Investigator, Massachusetts General Hospital
Other Study IDs: 2006P001624
Record Dates: First submitted 2008-12-02; First posted 2008-12-03 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2016-03

CONDITIONS: Neonatal Hyperbilirubinemia
MeSH Terms: conditions — Hyperbilirubinemia, Neonatal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Intervention: Receive decision support when reviewing bilirubin results in the clinical information systems/electronic health record
- Control: No decision support

SUMMARY:
We will use information technology to integrate the 2004 American Academy of Pediatrics guidelines for management of neonatal hyperbilirubinemia with laboratory reporting of newborn bilirubin test results to improve physician adherence to the guidelines and quality of care.

DETAILED DESCRIPTION:
In 2004, the American Academy of Pediatrics disseminated clinical practice guidelines for the management of neonatal hyperbilirubinemia. Using the infant's age in hours, serum bilirubin levels are applied to hour-specific nomograms to assess risk of developing significant hyperbilirubinemia as well as the necessity for treatment. Prior guidelines did not include nomograms for either. A systems approach to managing neonatal hyperbilirubinemia, including use of the nomograms, has been shown to improve outcomes and patient safety.

Despite the existence of these guidelines, decision support does not exist within MGH clinical information systems for managing neonatal hyperbilirubinemia. We propose to create BiliCurves, an application that integrates perinatal information from the obstetrical health record with that of the newborn's, providing seamless reporting of neonatal bilirubin results in the context of the practice guidelines and relevant obstetrical data. BiliCurves will graphically superimpose bilirubin results onto hour-specific guideline nomograms that providers can view when viewing bilirubin results. We propose to randomize BiliCurves access to pediatric providers, and study its effects on management of hyperbilirubinemia both during birth hospitalization as well as in the outpatient setting after discharge. We hypothesize infants treated by physicians with BiliCurves access will receive birth hospitalization phototherapy at a higher rate and readmission for hyperbilirubinemia at a lower rate than that of the control group. We also hypothesize that physicians with BiliCurves access will report greater ease and confidence in nomogram use and providing evidence-based care as BiliCurves obviates the provider having to have access to paper based versions of the nomogram (usual care) as well decreases potential errors in plotting test results on the nomograms.

ELIGIBILITY:
Inclusion Criteria:

* Providers who care for infants in the newborn nursery.
* All newborns in the newborn nursery that are 35 weeks or more weeks of gestation will be study eligible.

Exclusion Criteria:

* Infants less than 35 weeks gestation.

Max Age: 1 Month | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Providers who care for infants in the newborn nursery at MGH will be study eligible. All newborns 35 weeks or more weeks of gestation will be study eligible.
Sampling Method: Non-Probability Sample
Enrollment: 273 (Actual)
Dates: Start 2008-11; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Adherence to clinical guidelines | Initial Newborn Inpatient Stay, which on average is 2-3 days in length
  Adeherence to AAP clinical guidelines in treating neonatal hyperbilirubinemia

CONTACTS AND LOCATIONS:
Overall Officials: John Patrick T Co, MD, MPH, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] American Academy of Pediatrics Subcommittee on Hyperbilirubinemia. Management of hyperbilirubinemia in the newborn infant 35 or more weeks of gestation. Pediatrics. 2004 Jul;114(1):297-316. doi: 10.1542/peds.114.1.297. PMID 15231951